CLINICAL TRIAL: NCT01179685
Title: Diagnostic Utility of Pleural Fluid MAGE Assay in Patients With Pleural Effusion From Primary Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Institutional Review Board, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-08-043
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Unilatral Pleural Effusion

INTERVENTIONS:
Procedure: pleural fluid tapping — Minimally invasive technique to detect malignant pleural effusion

SUMMARY:
Melanoma antigen (MAGE) gene is known to be expressed in tumor cells, testis and placenta. The purpose of this prospective study was to investigate the sensitivity, specificity and accuracy of pleural fluid MAGE gene expression, tumor marker and cytology in the diagnosis of malignant pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* unilateral pleural effusion on chest radiography

Exclusion Criteria:

* body temperature > 38.3ºC and peripheral blood leukocytosis (>12,000/μl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The purpose of this prospective study was to investigate the sensitivity, specificity and accuracy of pleural fluid MAGE gene expression, tumor marker and cytology in the diagnosis of malignant pleural effusion. | 12months interval

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Won Um, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea